CLINICAL TRIAL: NCT04883021
Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation for Treatment of Methamphetamine Use Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of New Mexico (Other)
Collaborators: University of Iowa (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNM HRRC# 20-077
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-05

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Intervention Model Description: Single arm prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dual Target Theta Burst Stimulation (Experimental): The TMS intervention is open-label dual-target theta burst stimulation delivered in sequential fashion to the DLPFC and the MPFC.
  Interventions: Device: Dual Target Theta Burst Stimulation

INTERVENTIONS:
Device: Dual Target Theta Burst Stimulation — TMS treatment will be provided daily for 5 days, then daily for 5 days in week 2, and three times per week (Monday, Wednesday, Friday) in weeks 3 and 4.
  Treatment targeting will occur at the Beam F3 and FP1 scalp regions as defined by the 10-20 EEG system and previous publications. A Magventure MagPro X100 figure-8 coil with theta burst capabilities will be used to deliver the stimulus, including intermittent theta burst stimulation to the DLPFC (2 seconds of 50-Hz triplets delivered at 5 Hz, 8 seconds intertrain interval, 600 total pulses) and continuous theta burst to the MPFC (continuous 50-Hz stimulation triplets, 600 pulses). Stimulation will be delivered at 110% of the resting motor threshold.

SUMMARY:
We propose a single-arm clinical trial, with historical controls as a comparison group for select outcomes. Subjects with MAUD will receive 16 sessions of dual-target theta burst stimulation to the DLPFC and MPFC over 4 weeks. We will follow outcomes for 12 weeks. Outcomes include treatment retention, craving, self-reported MA or stimulant use, urine drug screen results, depressive symptoms, anxiety symptoms, sleep quality, quality of life, response inhibition, and functional connectivity. Magnetic resonance imaging (MRI) to measure functional connectivity at baseline and four weeks.

DETAILED DESCRIPTION:
Methamphetamine (MA) use can cause many serious adverse health consequences and is an important public health issue in Iowa, New Mexico, and Utah. In the 2017 Treatment Episode Data Set, 26% of substance use disorder treatment admissions from these states involved MA as the primary substance. MA-involved overdose deaths have been increasingly common in these states. Treatment for MA use disorder (MAUD) is primarily psychosocial. Rates of treatment induction and retention are poor, and relapse rates are high. There is a pressing need to identify effective interventions that enhance psychosocial treatments.

Transcranial magnetic stimulation (TMS) using either high frequency stimulation or intermittent theta burst stimulation is a non-invasive brain stimulation technique that effectively treats major depressive disorder and is considered safe, well-tolerated, and potent. TMS has increasingly been studied to treat addiction. The dorsolateral prefrontal cortex (DLPFC), a brain region implicated in regulatory processes related to executive function, emotion, motivation, and craving, is a common target for TMS. DLPFC stimulation using high frequency repetitive TMS has reduced craving in many studies of addictive disorders, including cocaine and MAUD. In addition to the DLPFC target, emerging evidence indicates that continuous theta burst stimulation (cTBS) delivered to the medial prefontal cortex (MPFC) during drug cue activation reduced craving and related brain activity in cocaine users. Despite these encouraging findings, no trials have reported on the efficacy of TMS for reducing MA use or preventing relapse. Clinical research on TMS for MAUD is sparse in the United States, and the limited studies of TMS in MAUD have been in experimental or closed treatment settings where effects on actual MA use are difficult to evaluate.

We are proposing a pilot study in 8 people with MAUD engaged in psychosocial treatment to explore the effects and tolerability of a four-week treatment protocol combining intermittent theta burst stimulation of the DLPFC with cTBS targeting the MPFC (dual-target TMS). We expect that this combined approach will enhance executive function and inhibitory control and reduce craving through separate but related mechanisms. We will evaluate clinical outcomes including symptoms and substance use, changes in functional connectivity measured via MRI and their relationship to treatment response, and changes in impulsivity as measured by performance on a response inhibition task. This project has the following specific aims:

Aim 1: Characterize changes in craving, depressive symptoms, anxiety symptoms, sleep quality, quality of life, and MA or other stimulant use over four weeks of dual-target TMS and eight weeks of subsequent follow-up.

Aim 2: Estimate changes in functional connectivity in the brain and response inhibition and selective attention in people with MAUD after four weeks of dual-target TMS.

Aim 3: Evaluate retention in the study to establish feasibility and tolerability of the protocol.

Aim 4: Compare retention in psychosocial treatment and positive urine drug screens in study participants compared to matched historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an active methamphetamine use disorder
* Is engaged in psychosocial treatment or articulates a plan to engage in psychosocial treatment for methamphetamine use disorder during the study period
* Age 18 to 60 years
* Able to consent for treatment and research participation
* English-speaking

Exclusion Criteria:

* Age less than 18 years (TMS not studied in pediatric population)
* Patients that are excluded during TMS assessment including: patients with epilepsy or seizure disorder, patients with implanted ferromagnetic equipment in their face or skull near the stimulation target.
* Current medical treatment with clozapine, bupropion, or stimulants.
* Current diagnosis of bipolar disorder, schizoaffective disorder, schizophrenia, or any other psychotic disorder.
* Legal or mental incompetency, or inability to consent to study.
* Unstable medical illness.
* Current diagnosis of neurological disorder or neurocognitive disorder.
* Prior neurosurgical procedure.
* History of seizure.
* History of ECT treatment within the past three months.
* History of any previous TMS treatment.
* Inability to complete the protocol, namely, inability to independently attend all study visits and TMS sessions on time.
* Prisoner
* Implanted device including pacemaker, coronary stent, defibrillator, or neurostimulation device that is not MRI-compatible
* Metal in body including bullets, shrapnel, metal slivers
* Claustrophobia
* Uncontrolled high blood pressure
* Atrial fibrillation
* Significant heart disease
* Hemodynamic instability
* Kidney disease
* Pregnant (MRI contraindicated during pregnancy)
* Unable to understand English (behavioral tests of impulsivity are only in English)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Rate of Retention in Study | 4 week visit
  Percentage of subjects who complete the 4-week TMS treatment period.
Change in functional connectivity | 4 week visit
  Change in connectivity index between the dorsolateral prefrontal cortex (DLPFC) and anterior insula
Change in Craving | 4 week visit
  Change in the Brief Substance Craving Scale Score

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No